CLINICAL TRIAL: NCT03036605
Title: The Postoperative Analgesic Effect of Dexamethasone Added to Topical Bupivacaine in Endoscopic Nasal Surgery
Brief Title: The Effect of Dexamethasone Added to Bupivacain in Nasal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ataturk University
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Nasal Surgery
Keywords: dexamethasone; bupivacaine; nasal surgery; nasal packing
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Bupivacaine (Active Comparator): 4 ml %0.5 bupivacaine and 1 ml %0.9 NaCl infiltration into nasal packing to both sides
  Interventions: Drug: Bupivacaine
- Group Bupivacaine+Dexamethasone (Active Comparator): 4 ml %0.5 bupivacaine and 4mg(1 ml) dexamethasone infiltration into nasal packing to both sides
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — %0.5 bupivacaine
  Other Names: Bupivacaine only
Drug: Dexamethasone — 8 mg Dexamethasone
  Other Names: Bupivacaine plus dexamethasone
  Arms: Group Bupivacaine+Dexamethasone

SUMMARY:
Nasal packing is frequently applied after nasal surgery. Nasal packing reduces epistaxis, prevents septal hematoma and stabilizes nasal septum. Nasal mucosa is quite sensitive to pain, therefore the most common problems after surgery are postoperative pain and anxiety during removal of the nasal packing. Lots of methods have been tried to control this pain (non-steroidal anti-inflammatory drugs, nerve blockade with long-acting local anesthetics, local anesthetics infiltration into nasal packing).

Glucocorticoids have been used as an adjuvant in the management of acute postoperative pain. Perineural dexamethasone as an adjuvant for the single-injection nerve block can prolong analgesia and reduce opioid-requiring after surgery. Furthermore dexamethasone reduces postoperative nausea and vomiting incidance.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients undergoing nasal surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | Postoperative 24 hours
  Analgesic consumption first 24 hours

SECONDARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively.
Visual analog pain score | postoperative second hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual analog pain score | postoperative 4th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively.
Visual analog pain score | postoperative 8th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively.
Visual analog pain score | postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Murat Yayik, MD, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sahin C, Aras HI. Effect on patient anxiety of lidocaine infiltration into nasal packing after septoplasty: prospective, controlled study. J Laryngol Otol. 2015 Aug;129(8):784-7. doi: 10.1017/S0022215115001644. Epub 2015 Jun 29. PMID 26118324
- [Background] Yilmaz S, Kocaman Akbay B, Yildizbas S, Guclu E, Yaman H, Yalcin Sezen G. Efficacy of topical levobupivacaine in control of postoperative pain after septoplasty. J Otolaryngol Head Neck Surg. 2010 Aug;39(4):454-7. PMID 20643015
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Bjorn S, Linde F, Nielsen KK, Borglum J, Hauritz RW, Bendtsen TF. Effect of Perineural Dexamethasone on the Duration of Single Injection Saphenous Nerve Block for Analgesia After Major Ankle Surgery: A Randomized, Controlled Study. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):210-216. doi: 10.1097/AAP.0000000000000538. PMID 28033159